CLINICAL TRIAL: NCT03383757
Title: U-TruSignal SpO2 Testing in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 123.04-2017-GES-0002
Record Dates: First submitted 2017-11-03; First posted 2017-12-26 (Actual); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Pulse Oximetry
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SpO2 Sensor Application & Blood draw (Experimental): All subjects will undergo the same study procedures of having their SpO2 levels measured with an external sensor applied to the skin and blood SpO2 level measured
  Interventions: Device: SpO2 Sensor application & blood draw

INTERVENTIONS:
Device: SpO2 Sensor application & blood draw — At the start of the procedure, one to two commercial sensors shall be applied to the subject. Readings will be allowed to stabilize. After at least 10 minutes of data collection, arterial blood will be collected and analyzed blood per hospital's standard procedure. Data collection will continue post blood draw for two minutes.

SUMMARY:
The purpose of the study is to demonstrate proper function of the U-TruSignal device via clinical performance testing in a neonatal human subject population under standard clinical conditions. A study with human subjects will provide the needed clinical evidence for assessing the accuracy of the pulse oximeter as recommended by the FDA Guidance Document (Pulse Oximeters - Premarket Notification Submissions [50(k)s]: Guidance for Industry and Food and Drug Administration Staff.)

DETAILED DESCRIPTION:
The purpose of this study is to collect blood samples from neonates under normal clinical conditions to ensure proper function (clinical performance) with the U-TruSignal device.

The study will include both the TruSignal AllFit Sensor and TruSignal Sensitive Sensor.

After providing consent, no preparation beyond the investigational site's standard of care is required before study procedures begin. At the start of the procedure, one to two sensors, upon the discretion of the investigator, shall be applied to the subject.

The duration of the subject's participation in the study is dependent upon the scheduled routine arterial blood draw and obtaining the maximum of 6 data pairs (3 data pairs per sensor). The Investigator or designated study staff will collect of SpO2 and pulse rate for each study subject. Laboratory results from arterial blood draw will be collected from the hospital's medical records. The description, severity, and device relatedness of any AE or SAE during the study will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Parents or legally authorized representative (LAR) can understand and provide written informed consent; AND
2. Subjects are < 29 days old, and requiring arterial blood samples per the site's standard of care.

Exclusion Criteria:

1. Neonates with injuries, deformities or abnormalities may prevent proper application of the sensor;
2. Neonates with inadequate heart pump function affecting blood circulation caused by identified cardiac or cardiovascular conditions such as patent ductus arteriosus, persistent pulmonary hypertension, septal defects, or congenital heart disease;
3. Neonates with mean arterial blood pressure < 20mmHg;
4. Neonates with congenital diaphragmatic hernia; OR
5. Neonates under High frequency ventilation therapy.

Max Age: 29 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Agarwal, MD, Principal Investigator — NH Narayana Multispecialty Hospital, Unit of Narayana Health, Mazumdar Shaw Medical Center; Outi Tammela, MD, Principal Investigator — Tampere University Hospital (TAYS)
Locations (2):
- Tampere University Hospital (TAYS), Tampere, Finland
- NH Narayana Multispecialty Hospital, Unit of Narayana Health, Mazumdar Shaw Medical Center, Bangalore, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SpO2 Sensor Application & Blood Draw: All subjects will undergo the same study procedures of having their SpO2 levels measured with an external sensor applied to the skin and blood SpO2 level measured. Subject may have one or both sensors applied.
  SpO2 Sensor application & blood draw: At the start of the procedure, one to two commercial sensors shall be applied to the subject. Readings will be allowed to stabilize. After at least 10 minutes of data collection, arterial blood will be collected and analyzed blood per hospital's standard procedure. Data collection will continue post blood draw for two minutes.
Period: Overall Study
Arm/Group | SpO2 Sensor Application & Blood Draw
Started | 117
TruSignal AllFit Sensor Subjects | 56
TruSignal Sensitive Sensor Subjects | 59
TruSignal AllFit Sensor Data Pairs | 52
TruSignal Sensitive Sensor Data Pairs | 51
Completed | 78
Not Completed | 39

BASELINE CHARACTERISTICS:
Arm/Group | SpO2 Sensor Application & Blood Draw
Number analyzed (Participants) | 78
Age, Customized [Mean (Standard Deviation); unit: days]
  Age | 5.2 (4.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Accuracy Root Mean Square (ARMS) Per Data Pair
Description: Compare observations of Peripheral Capillary Oxygen Saturation (SpO2- measured by the test pulse oximeter system) and Oxygen Saturation of Arterial Blood (SaO2) values (measured by CO-Oximeter analysis of simultaneous drawn arterial blood).
Time Frame: 30 minutes per data pair
Population: Participants may have multiple data points with multiple sensors.
Measure: Number; unit: percentage of oxygen saturated hemoglobi
Arm/Group | SpO2 Sensor Application & Blood Draw
Number analyzed (Participants) | 78
percentage of oxygen saturated hemoglobi
  TS-AF ARMS: number analyzed (Participants) | 38
  TS-AF ARMS | 2.57
  TS-SE ARMS: number analyzed (Participants) | 40
  TS-SE ARMS | 2.57

2. Secondary Outcome: Continuous SpO2 Measurements During Data Collection Interval
Description: The secondary objective of the study was to demonstrate U-TruSignal collects substantially continuous SpO2 measurements during a data collection interval. All time the sensors were worn and data collected across participants were reviewed for invalid data within each data pair. For the data pairs that had moments of invalid data, a calculation was conducted (invalid data/complete data for data pair) to establish percentage of invalid data per sensor. For each sensor type the percentage of invalid data (%) was calculated. Sensor readings were grouped together across participants and are being reported as the total number of invalid readings over the total number of readings for all participants
Time Frame: 30 minutes per data pair
Population: 78 Participants analyzed, 38 with TS-AF sensor, 40 with TS-SE sensor. Participants may have multiple data points with multiple sensors.
Measure: Count of Participants; unit: Participants
Arm/Group | SpO2 Sensor Application & Blood Draw
Number analyzed (Participants) | 78
Participants
  TS-AF <=1% of invalid data: number analyzed (Participants) | 38
  TS-AF <=1% of invalid data | 38
  TS-AF >1% of invalid data: number analyzed (Participants) | 38
  TS-AF >1% of invalid data | 0
  TS-SE <=1% of invalid data: number analyzed (Participants) | 40
  TS-SE <=1% of invalid data | 40
  TS-SE >1% of invalid data: number analyzed (Participants) | 40
  TS-SE >1% of invalid data | 0

3. Other Pre Specified Outcome: Type and Number of AEs, SAEs, and Device Issues
Description: Collect safety information, including type and number of AE s, SAEs, and device issues.
Time Frame: 30 minutes per data pair
Population: AE, SAE and Device Issues were measured for each sensor.
Measure: Number; unit: Events
Arm/Group | SpO2 Sensor Application & Blood Draw
Number analyzed (Participants) | 78
Events
  TruSignal AllFit Sensor AE: number analyzed (Participants) | 38
  TruSignal AllFit Sensor AE | 0
  TruSignal AllFit Sensor SAE: number analyzed (Participants) | 38
  TruSignal AllFit Sensor SAE | 0
  TruSignal AllFit Sensor Device Issues: number analyzed (Participants) | 38
  TruSignal AllFit Sensor Device Issues | 0
  TruSignal Sensitive Sensor AE: number analyzed (Participants) | 40
  TruSignal Sensitive Sensor AE | 0
  TruSignal Sensitive Sensor SAE: number analyzed (Participants) | 40
  TruSignal Sensitive Sensor SAE | 0
  TruSignal Sensitive Sensor Device Issues: number analyzed (Participants) | 40
  TruSignal Sensitive Sensor Device Issues | 0

ADVERSE EVENTS:
Time Frame: 1 hour.
Arm/Group | SpO2 Sensor Application & Blood Draw
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT03383757/Prot_SAP_000.pdf